CLINICAL TRIAL: NCT02438124
Title: Rhythmic Auditory Stimulation Optimalization for Gait Improvement in Parkinson's
Brief Title: Rhythmic Auditory Stimulation Optimalization for Gait Improvement in Parkinson's Disease - BeatPark Study
Acronym: BeatPark
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Université Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 9193-2
Record Dates: First submitted 2015-04-30; First posted 2015-05-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Rhythmic auditory stimulation; Gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient (Experimental): Patient with Parkinson's Disease with walking test and neuropsychological evaluation
  Interventions: Behavioral: Neuropsychological evaluation
- Contrôle (Experimental): normal control with walking test and neuropsychological evaluation
  Interventions: Behavioral: Neuropsychological evaluation

INTERVENTIONS:
Behavioral: Neuropsychological evaluation — The subjects are submitted in one hearing stimulus while they realize a walking test

SUMMARY:
The beneficial effects of rhythmical auditory stimulation (RAS) on spatio-temporal gait characteristics in Parkinson's disease (PD) are attested by clinical research.

Nonetheless, it is still unclear which auditory information parameters (i.e. complexity, temporal regularity or adaptability to gait) maximize the effectiveness of RAS.

Objectives: To evaluate the beneficial effects of RAS on spatio-temporal gait characteristics in PD patients with gait disorders according to:

* RAS complexity (i.e. metronome, amplitude modulated noise, music)
* RAS variability (i.e fixed, random, semi-random)
* RAS adapted in real-time to gait

Variability study:

To study the impact of RAS variability (i.e fixed, random, semi-random) in 20 PD patients and 20 healthy controls on spatio-temporal gait characteristics with metronome, amplitude noise and music.

Adaptability studyTo study the impact of RAS adaptability (i.e fixed, random, adapted in real-time to gait) in 20 PD patients and 20 healthy controls on spatio-temporal gait characteristics with metronome, amplitude noise and music.

ELIGIBILITY:
Inclusion Criteria:

* 18 y.o.
* to be able to understand the study aims and to agree to participate
* to have signed the consent form
* to be registered to social security system
* to reach the diagnosis criteria of idiopathic PD (Queen Square Brain Bank)
* gait disorder clinically observable

Exclusion Criteria:

* pregnant or lactating woman
* high probability of non-compliance
* curators , authorship or advisers to person of full age Specific exclusion criteria for PD patients
* clinical signs of parkinsonian syndrome
* Mini Mental State Examination < 24/30 Specific exclusion criteria for controls
* neurological disease
* gait disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-03 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
gait velocity | 2 days
  evaluation of walking speed between the different conditions

SECONDARY OUTCOMES:
spatio-temporal gait characteristics | 2 days
  evaluation of other walking parameters between the different conditions

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Cochen De Cock, MD, Principal Investigator — University Hospital, Montpellier
Locations (3):
- France (3):
  - Service de neurologie de la Clinique Beau Soleil, Montpellier
  - CIC, Montpellier
  - Plateau Technique de Rééducation Fonctionnelle (Hôpital Gui de Chauliac) du, Montpellier

REFERENCES:
- [Result] Arias P, Cudeiro J. Effects of rhythmic sensory stimulation (auditory, visual) on gait in Parkinson's disease patients. Exp Brain Res. 2008 Apr;186(4):589-601. doi: 10.1007/s00221-007-1263-y. Epub 2008 Jan 23. PMID 18214453
- [Result] Arias P, Cudeiro J. Effect of rhythmic auditory stimulation on gait in Parkinsonian patients with and without freezing of gait. PLoS One. 2010 Mar 22;5(3):e9675. doi: 10.1371/journal.pone.0009675. PMID 20339591
- [Result] Blin O, Ferrandez AM, Pailhous J, Serratrice G. Dopa-sensitive and dopa-resistant gait parameters in Parkinson's disease. J Neurol Sci. 1991 May;103(1):51-4. doi: 10.1016/0022-510x(91)90283-d. PMID 1865232
- [Result] Bloem BR, Hausdorff JM, Visser JE, Giladi N. Falls and freezing of gait in Parkinson's disease: a review of two interconnected, episodic phenomena. Mov Disord. 2004 Aug;19(8):871-84. doi: 10.1002/mds.20115. PMID 15300651
- [Result] Brown LA, de Bruin N, Doan JB, Suchowersky O, Hu B. Novel challenges to gait in Parkinson's disease: the effect of concurrent music in single- and dual-task contexts. Arch Phys Med Rehabil. 2009 Sep;90(9):1578-83. doi: 10.1016/j.apmr.2009.03.009. PMID 19735787
- [Result] Delignieres D, Torre K. Fractal dynamics of human gait: a reassessment of the 1996 data of Hausdorff et al. J Appl Physiol (1985). 2009 Apr;106(4):1272-9. doi: 10.1152/japplphysiol.90757.2008. Epub 2009 Feb 19. PMID 19228991
- [Result] Dujardin K, Sockeel P, Carette AS, Delliaux M, Defebvre L. Assessing apathy in everyday clinical practice with the short-form Lille Apathy Rating Scale. Mov Disord. 2013 Dec;28(14):2014-9. doi: 10.1002/mds.25584. Epub 2013 Jul 8. PMID 23836341
- [Result] Ebersbach G, Heijmenberg M, Kindermann L, Trottenberg T, Wissel J, Poewe W. Interference of rhythmic constraint on gait in healthy subjects and patients with early Parkinson's disease: evidence for impaired locomotor pattern generation in early Parkinson's disease. Mov Disord. 1999 Jul;14(4):619-25. doi: 10.1002/1531-8257(199907)14:43.0.co;2-x. PMID 10435499
- [Result] Elbers RG, van Wegen EE, Verhoef J, Kwakkel G. Is gait speed a valid measure to predict community ambulation in patients with Parkinson's disease? J Rehabil Med. 2013 Apr;45(4):370-5. doi: 10.2340/16501977-1123. PMID 23450464
- [Result] Gibb WR, Lees AJ. The relevance of the Lewy body to the pathogenesis of idiopathic Parkinson's disease. J Neurol Neurosurg Psychiatry. 1988 Jun;51(6):745-52. doi: 10.1136/jnnp.51.6.745. PMID 2841426
- [Result] Godefroy O, Brigitte A, Philippe A, Mira DH, Olivier G, Didier le G, Rose-Marie M, Thierry M, Chrystele M, Blandine P, Bernard P, Philippe R; Groupe de Reflexion sur L'Evaluation des Fonctions EXecutives. [Frontal dysexecutive syndromes]. Rev Neurol (Paris). 2004 Oct;160(10):899-909. doi: 10.1016/s0035-3787(04)71071-1. French. PMID 15492716
- [Result] Hausdorff JM. Gait dynamics in Parkinson's disease: common and distinct behavior among stride length, gait variability, and fractal-like scaling. Chaos. 2009 Jun;19(2):026113. doi: 10.1063/1.3147408. PMID 19566273
- [Result] Hove MJ, Suzuki K, Uchitomi H, Orimo S, Miyake Y. Interactive rhythmic auditory stimulation reinstates natural 1/f timing in gait of Parkinson's patients. PLoS One. 2012;7(3):e32600. doi: 10.1371/journal.pone.0032600. Epub 2012 Mar 2. PMID 22396783
- [Result] Howe TE, Lovgreen B, Cody FW, Ashton VJ, Oldham JA. Auditory cues can modify the gait of persons with early-stage Parkinson's disease: a method for enhancing parkinsonian walking performance? Clin Rehabil. 2003 Jul;17(4):363-7. doi: 10.1191/0269215503cr621oa. PMID 12785243
- [Result] Hughes AJ, Daniel SE, Kilford L, Lees AJ. Accuracy of clinical diagnosis of idiopathic Parkinson's disease: a clinico-pathological study of 100 cases. J Neurol Neurosurg Psychiatry. 1992 Mar;55(3):181-4. doi: 10.1136/jnnp.55.3.181. PMID 1564476
- [Result] Judge JO, Davis RB 3rd, Ounpuu S. Step length reductions in advanced age: the role of ankle and hip kinetics. J Gerontol A Biol Sci Med Sci. 1996 Nov;51(6):M303-12. doi: 10.1093/gerona/51a.6.m303. PMID 8914503
- [Result] Kerr GK, Worringham CJ, Cole MH, Lacherez PF, Wood JM, Silburn PA. Predictors of future falls in Parkinson disease. Neurology. 2010 Jul 13;75(2):116-24. doi: 10.1212/WNL.0b013e3181e7b688. Epub 2010 Jun 23. PMID 20574039
- [Result] Kirschner S, Tomasello M. Joint drumming: social context facilitates synchronization in preschool children. J Exp Child Psychol. 2009 Mar;102(3):299-314. doi: 10.1016/j.jecp.2008.07.005. Epub 2008 Sep 12. PMID 18789454
- [Result] Lehman DA, Toole T, Lofald D, Hirsch MA. Training with verbal instructional cues results in near-term improvement of gait in people with Parkinson disease. J Neurol Phys Ther. 2005 Mar;29(1):2-8. doi: 10.1097/01.npt.0000282256.36208.cf. PMID 16386155
- [Result] Lim I, van Wegen E, de Goede C, Deutekom M, Nieuwboer A, Willems A, Jones D, Rochester L, Kwakkel G. Effects of external rhythmical cueing on gait in patients with Parkinson's disease: a systematic review. Clin Rehabil. 2005 Oct;19(7):695-713. doi: 10.1191/0269215505cr906oa. PMID 16250189
- [Result] Marchese R, Diverio M, Zucchi F, Lentino C, Abbruzzese G. The role of sensory cues in the rehabilitation of parkinsonian patients: a comparison of two physical therapy protocols. Mov Disord. 2000 Sep;15(5):879-83. doi: 10.1002/1531-8257(200009)15:53.0.co;2-9. PMID 11009194
- [Result] Marmelat V, Delignieres D. Strong anticipation: complexity matching in interpersonal coordination. Exp Brain Res. 2012 Oct;222(1-2):137-48. doi: 10.1007/s00221-012-3202-9. Epub 2012 Aug 4. PMID 22865163
- [Result] McIntosh GC, Brown SH, Rice RR, Thaut MH. Rhythmic auditory-motor facilitation of gait patterns in patients with Parkinson's disease. J Neurol Neurosurg Psychiatry. 1997 Jan;62(1):22-6. doi: 10.1136/jnnp.62.1.22. PMID 9010395
- [Result] McIntosh, G.C., Rice, R.R., Hurt, C.P., and Thaut, M.H. (1998). Long-term training effects of rhythmic auditory stimulation on gait in patients with Parkinson's disease. Mov. Disord. Off. J. Mov. Disord. Soc. 13 (supple2), 212.
- [Result] Muslimovic D, Post B, Speelman JD, Schmand B, de Haan RJ; CARPA Study Group. Determinants of disability and quality of life in mild to moderate Parkinson disease. Neurology. 2008 Jun 3;70(23):2241-7. doi: 10.1212/01.wnl.0000313835.33830.80. PMID 18519873
- [Result] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Result] Nieuwboer A. Cueing for freezing of gait in patients with Parkinson's disease: a rehabilitation perspective. Mov Disord. 2008;23 Suppl 2:S475-81. doi: 10.1002/mds.21978. PMID 18668619
- [Result] Nieuwboer A, Kwakkel G, Rochester L, Jones D, van Wegen E, Willems AM, Chavret F, Hetherington V, Baker K, Lim I. Cueing training in the home improves gait-related mobility in Parkinson's disease: the RESCUE trial. J Neurol Neurosurg Psychiatry. 2007 Feb;78(2):134-40. doi: 10.1136/jnnp.200X.097923. PMID 17229744
- [Result] Nombela C, Hughes LE, Owen AM, Grahn JA. Into the groove: can rhythm influence Parkinson's disease? Neurosci Biobehav Rev. 2013 Dec;37(10 Pt 2):2564-70. doi: 10.1016/j.neubiorev.2013.08.003. Epub 2013 Sep 3. PMID 24012774
- [Result] del Olmo MF, Cudeiro J. Temporal variability of gait in Parkinson disease: effects of a rehabilitation programme based on rhythmic sound cues. Parkinsonism Relat Disord. 2005 Jan;11(1):25-33. doi: 10.1016/j.parkreldis.2004.09.002. Epub 2004 Dec 9. PMID 15619459
- [Result] Post B, Muslimovic D, van Geloven N, Speelman JD, Schmand B, de Haan RJ; CARPA-study group. Progression and prognostic factors of motor impairment, disability and quality of life in newly diagnosed Parkinson's disease. Mov Disord. 2011 Feb 15;26(3):449-56. doi: 10.1002/mds.23467. Epub 2011 Feb 10. PMID 21312273
- [Result] Rascol O, Goetz C, Koller W, Poewe W, Sampaio C. Treatment interventions for Parkinson's disease: an evidence based assessment. Lancet. 2002 May 4;359(9317):1589-98. doi: 10.1016/S0140-6736(02)08520-3. PMID 12047983
- [Result] Repp BH. Sensorimotor synchronization: a review of the tapping literature. Psychon Bull Rev. 2005 Dec;12(6):969-92. doi: 10.3758/bf03206433. PMID 16615317
- [Result] Repp BH, Su YH. Sensorimotor synchronization: a review of recent research (2006-2012). Psychon Bull Rev. 2013 Jun;20(3):403-52. doi: 10.3758/s13423-012-0371-2. PMID 23397235
- [Result] Rizzolatti G, Fogassi L, Gallese V. Neurophysiological mechanisms underlying the understanding and imitation of action. Nat Rev Neurosci. 2001 Sep;2(9):661-70. doi: 10.1038/35090060. No abstract available. PMID 11533734
- [Result] Schaafsma JD, Giladi N, Balash Y, Bartels AL, Gurevich T, Hausdorff JM. Gait dynamics in Parkinson's disease: relationship to Parkinsonian features, falls and response to levodopa. J Neurol Sci. 2003 Aug 15;212(1-2):47-53. doi: 10.1016/s0022-510x(03)00104-7. PMID 12809998
- [Result] Sowinski J, Dalla Bella S. Poor synchronization to the beat may result from deficient auditory-motor mapping. Neuropsychologia. 2013 Aug;51(10):1952-63. doi: 10.1016/j.neuropsychologia.2013.06.027. Epub 2013 Jul 6. PMID 23838002
- [Result] Spaulding SJ, Barber B, Colby M, Cormack B, Mick T, Jenkins ME. Cueing and gait improvement among people with Parkinson's disease: a meta-analysis. Arch Phys Med Rehabil. 2013 Mar;94(3):562-70. doi: 10.1016/j.apmr.2012.10.026. Epub 2012 Nov 2. PMID 23127307
- [Result] Studenski S, Perera S, Patel K, Rosano C, Faulkner K, Inzitari M, Brach J, Chandler J, Cawthon P, Connor EB, Nevitt M, Visser M, Kritchevsky S, Badinelli S, Harris T, Newman AB, Cauley J, Ferrucci L, Guralnik J. Gait speed and survival in older adults. JAMA. 2011 Jan 5;305(1):50-8. doi: 10.1001/jama.2010.1923. PMID 21205966
- [Result] Thaut MH, McIntosh GC, Rice RR, Miller RA, Rathbun J, Brault JM. Rhythmic auditory stimulation in gait training for Parkinson's disease patients. Mov Disord. 1996 Mar;11(2):193-200. doi: 10.1002/mds.870110213. PMID 8684391
- [Result] Thaut MH, McIntosh KW, McIntosh GC, Hoemberg V. Auditory rhythmicity enhances movement and speech motor control in patients with Parkinson's disease. Funct Neurol. 2001 Apr-Jun;16(2):163-72. No abstract available. PMID 11495422
- [Result] Vu TC, Nutt JG, Holford NH. Progression of motor and nonmotor features of Parkinson's disease and their response to treatment. Br J Clin Pharmacol. 2012 Aug;74(2):267-83. doi: 10.1111/j.1365-2125.2012.04192.x. PMID 22283961
- [Result] Willems AM, Nieuwboer A, Chavret F, Desloovere K, Dom R, Rochester L, Jones D, Kwakkel G, Van Wegen E. The use of rhythmic auditory cues to influence gait in patients with Parkinson's disease, the differential effect for freezers and non-freezers, an explorative study. Disabil Rehabil. 2006 Jun 15;28(11):721-8. doi: 10.1080/09638280500386569. PMID 16809215
- [Result] Wright WG, Gurfinkel VS, King LA, Nutt JG, Cordo PJ, Horak FB. Axial kinesthesia is impaired in Parkinson's disease: effects of levodopa. Exp Neurol. 2010 Sep;225(1):202-9. doi: 10.1016/j.expneurol.2010.06.016. Epub 2010 Jul 1. PMID 20599976
- [Result] Yardley L, Beyer N, Hauer K, Kempen G, Piot-Ziegler C, Todd C. Development and initial validation of the Falls Efficacy Scale-International (FES-I). Age Ageing. 2005 Nov;34(6):614-9. doi: 10.1093/ageing/afi196. PMID 16267188
- [Result] Zatorre RJ, Chen JL, Penhune VB. When the brain plays music: auditory-motor interactions in music perception and production. Nat Rev Neurosci. 2007 Jul;8(7):547-58. doi: 10.1038/nrn2152. PMID 17585307
- [Result] Zentner M, Eerola T. Rhythmic engagement with music in infancy. Proc Natl Acad Sci U S A. 2010 Mar 30;107(13):5768-73. doi: 10.1073/pnas.1000121107. Epub 2010 Mar 15. PMID 20231438